CLINICAL TRIAL: NCT02487940
Title: Assessment of the Efficacy of Intralipid 20% in Management of Women With Unexplained Recurrent Implantation Failure in IVF Cycles: A Double Blinded Randomised Controlled Trial
Brief Title: Assessment of Intralipid Efficacy in Women With Unexplained Recurrent Implantation Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dar El Teb Institute (Other)
Responsible Party: Principal Investigator, ISLAM GAMALELDIN, Specialist registrar Obstetrics and Gynaecology, Dar El Teb Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASUH1234
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Subfertility
Keywords: Recurrent implantation failure; IVF; ICSI; Intralipid
MeSH Terms: conditions — Infertility | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intralipid (Active Comparator): Women with RIF received intralipid 20% (at a dose of 9mg/mL of the total blood volume, corresponding to 2 mL intralipid diluted at 20% in 250 mL normal saline) given over 1-2 hours on the day of oocyte retrieval. Dose is repeated on/the following day of a positive pregnancy test, followed by a final dose 2-3 weeks later when attending for pregnancy scan.
  Interventions: Drug: Intralipid 20%
- Placebo (Placebo Comparator): Women with RIF received intravenous infusion of 250 mL physiological saline solution over 1-2 hours on the day of oocyte retrieval. Dose is repeated on/the following day of a positive pregnancy test, followed by a final dose 2-3 weeks later when attending for pregnancy scan.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Intralipid 20% — Women with RIF received intralipid 20% (at a dose of 9mg/mL of the total blood volume, corresponding to 2 mL intralipid diluted at 20% in 250 mL normal saline) given over 1-2 hours on the day of oocyte retrieval. Dose is repeated on/the following day of a positive pregnancy test, followed by a final dose 2-3 weeks later when attending for pregnancy scan.
  Other Names: Lipofundin 20%
  Arms: Intralipid
Drug: Normal saline — Women with RIF received intravenous infusion of 250 mL physiological saline solution over 1-2 hours on the day of oocyte retrieval. Dose is repeated on/the following day of a positive pregnancy test, followed by a final dose 2-3 weeks later when attending for pregnancy scan.
  Other Names: Solution of sodium chloride
  Arms: Placebo

SUMMARY:
The study will include 100 women with unexplained recurrent implantation failure undergoing IVF/ICSI cycle.

Patients fulfilling the inclusion criteria will be randomised into two groups.

Study Group:

This group will include 50 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of intralipid 20%, on the day of oocyte retrieval, a second dose on/ the following day of positive pregnancy test and a final dose 2-3 weeks later when attending for pregnancy scan.

Control Group:

This group will include 50 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of placebo, on the day of oocyte retrieval, a second dose on/ the following day of positive pregnancy test and a final dose 2-3 weeks later when attending for pregnancy scan.

DETAILED DESCRIPTION:
The study will include 100 women with unexplained recurrent implantation failure undergoing IVF/ICSI cycle.

Randomisation:

Patients fulfilling the inclusion criteria will randomised to two groups.

Study Group:

This group will include 50 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of intralipid 20%, on the day of oocyte retrieval, a second dose on/ the following day of positive pregnancy test and a final dose 2-3 weeks later when attending for pregnancy scan.

Control Group:

This group will include 50 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of placebo, on the day of oocyte retrieval, a second dose on/ the following day of positive pregnancy test and a final dose 2-3 weeks later when attending for pregnancy scan.

Random allocation sequence generation:

A computer generated list will be used, assigning each participant number to either study groups.

Allocation Concealment:

Assignment will be done by sequentially numbered, otherwise identical, sealed envelopes (SNOSE), each containing a 2-inch by 2-inch paper with a written code designating the assigned group. These papers will be placed in a folded sheet of aluminium foil fitted inside the envelope. Effort will be taken to assure absence of any detectable differences in size or weight between intervention and control envelopes. Envelopes will be chosen to be opaque and lined inside with carbon paper. Envelopes will be opened sequentially only after writing the subject's tracking information on the envelope so that the carbon paper served as an audit trail.

Blinding:

Both drug with active ingredient and placebo will be provided by the hospital pharmacy in identical sealed opaque containers, equal in weight, similar in appearance, and tamper-proof. The drug with the active ingredient containers will be labeled either Group A or Group B by the head pharmacist and the assignment kept secret to be revealed after the end of the study.

Drugs will be administered to patients by a sealed opaque infusion drip.

IVF/ICSI cycle will be done using the standard LLP in both groups.

Primary outcome will be Live birth rates.

Secondary outcomes will be clinical pregnancy rates and side effects/tolerability of Intralipid infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-38 years of age.
* Repeated implantation failure with 3 or more failed IVF cycles with good quality embryos.
* Normal trans-vaginal ultrasonography.
* Normal hysteroscopy.
* Normal male and female karyotyping.
* Normal anti cardiolipin antibody IGG, IGM and Lupus anticoagulant.
* Normal thrombophilia screen in the form of protein c, s, anti thrombin iii and factor v leiden.
* Written and signed informed consent by the patient to participate in the study.

Exclusion Criteria:

* Age more than 38 years.
* Less than 3 failed IVF cycles.
* Poor embryo quality.
* Expected poor ovarian response.
* Abnormal trans-vaginal ultrasound findings e.g. endometrial polyps or fibroids.
* Abnormal male or female karyotyping.
* Abnormal hysteroscopic finding e.g. endometrial polyps, endometrial hyperplasia, fibroid or congenital anomalies.
* Positive Anticardiolipin antibodies or Lupus anticoagulant.
* Positive thrombophilia screen.
* Allergy to soy oil, eggs, peanut, peanut-based products or any active ingredient in the infusion.
* Mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Live birth rates | up to 40 weeks gestation

SECONDARY OUTCOMES:
Clinical pregnancy rates | 6 weeks gestation (2 weeks following embryo transfer)
side effects and tolerability of Intralipid | up to 40 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Gomaa, MD, Study Director — Ain Shams univeristy hospitals

IPD SHARING:
Plan to Share IPD: Yes